CLINICAL TRIAL: NCT05838677
Title: Multicentre Pragmatic Cluster Randomised Controlled Feasibility Trial to Assess Potential Effectiveness and Cost-effectiveness of the Pain at Work Toolkit in Employees With Chronic or Persistent Pain
Brief Title: Pain at Work Toolkit in Employees With Chronic Pain
Acronym: PAW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nuffield Trust (Unknown); University of Aberdeen (Other); University of Exeter (Other); Monash University (Other); Versus Arthritis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Blake_PAWFeasibilityTrial_2023; DERR1-10.2196/51474 (Registry Identifier: International Registered Report Identifier (IRRID)); OBF/FR-000023820 (Other Grant/Funding Number: NNuffield Foundation's Oliver Bird Fund and Versus Arthritis)
Record Dates: First submitted 2023-03-27; First posted 2023-05-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain; Pain, Chronic
MeSH Terms: conditions — Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This study is an open-label, two-arm, multicentre, pragmatic cluster randomised controlled feasibility trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Pain at Work Toolkit (Experimental): Intervention participants receive the PAW toolkit plus 3 x optional occupational therapy calls (approximately 30 minutes each) involving orientation to the PAW Toolkit and individually tailored advice and behavioural strategies for managing pain at work. This digital web-based toolkit is designed to support people with chronic pain in self-managing their condition at work. PAW offers evidence-based advice about chronic or persistent pain, disability rights, work capacity, pain self-management strategies and signposting to support.
  Interventions: Behavioral: Pain at Work Toolkit
- Active Control Group: Treatment as Usual (Active Comparator): Participants do not receive the PAW Toolkit but instead have treatment as usual (TAU) from their employer. The nature of TAU will be recorded as part of the feasibility study. Depending on the employing organisation, TAU may consist of (but is not limited to) any combination of the following: occupational health, counselling, line manager support, signposting to education about factors that may have positive or negative effects on chronic pain. Participants can access non-specialist telephone calls from a researcher to discuss their participation in the study.
  Interventions: Other: Active control

INTERVENTIONS:
Behavioral: Pain at Work Toolkit — Online toolkit providing advice and signposting to help people self-manage chronic or persistent pain at work. Access to optional phone call support from an occupational therapist providing individually tailored advice.
  Other Names: PAW Toolkit
  Arms: Intervention Group: Pain at Work Toolkit
Other: Active control — Treatment as usual which will vary depending on the employing organisation but may include, for example, line manager support, occupational health input etc. Access to optional non-specialist phone call support from a study researcher.
  Other Names: Treatment as usual (TAU)
  Arms: Active Control Group: Treatment as Usual

SUMMARY:
This project will test the feasibility and acceptability of the Pain at Work (PAW) Toolkit which aims to help employees self-manage chronic or persistent pain at work. Ultimately, the investigators want to discover if it improves employees' health, wellbeing, confidence to self-manage their condition, and reduces impacts on their ability to work and be productive at work. Prior to testing the effectiveness and cost-effectiveness of the PAW Toolkit in a large-scale randomised trial, the investigators are conducting a multicentre pragmatic cluster randomised controlled feasibility trial. This will establish whether the PAW Toolkit, and our research processes, are feasible and acceptable in workplace settings, and will inform the design of a future trial. In this feasibility study, organisations will be randomised at site level to receive the intervention (PAW Toolkit plus occupational therapist (OT) support calls) or control (treatment as usual) for any individual employees who consent to take part. The investigators aim to recruit around 120 participants ("individual employees") from around 8 sites ("clusters"). Data will be collected from employees and organisations at baseline, 3 months and 6 months, using online surveys. At 6 months, up tp 40 people from across different sites and job roles will be interviewed, including employees who have accessed the PAW Toolkit, and other stakeholders (people who have been involved in supporting them at work, such as their line manager).

The data will be used assess whether the intervention and the research processes are acceptable and feasible, and the information collected will be used to plan a large-scale randomised controlled trial.

DETAILED DESCRIPTION:
Background:

Chronic or persistent pain affects around 28 million adults in the United Kingdom (UK), reducing quality of life and people's ability to work or be productive at work. Sickness absence and reduced productivity costs the UK economy £73 billion per year.

Access to work advice and support for people living with pain is variable. Most people with chronic pain do not receive work advice through healthcare services, and employers do not routinely provide education or support for people with chronic pain. The Pain at Work (PAW) Toolkit aims to equip people who have pain with the knowledge, skills and confidence to: effectively self-manage a painful condition at work; access help and support; enjoy a better work experience; remain in the workforce.

Aims:

The aim of the trial is to determine the feasibility of conducting a definitive cluster randomised controlled trial (cRCT) of the effectiveness and cost-effectiveness of the PAW Toolkit for working-age adults with chronic or persistent pain. To achieve this, the objectives are:

* To measure feasibility outcomes to assess whether it would be possible to recruit to a definitive trial (recruitment, retention).
* To test the feasibility of reaching different employee groups (e.g., age, gender, ethnicity, job role or type), sectors (e.g., public, private, third) and organisation types (e.g., small-to-medium, or large enterprises).
* To explore whether participants and employers find the intervention and trial design acceptable.
* To obtain an estimate of the intra-cluster correlation coefficient to inform the future sample size calculation for the main trial.
* To collect a range of outcome measures to help identify the most appropriate primary outcome for a definitive trial.
* To collect data to assess the feasibility of capturing health economic data in a future trial.
* To design a future trial and implementation plan.

Protocol/ Method:

Trial configuration includes 3 work packages (WP's): feasibility trial (WP1); health economics evaluation (WP2); nested interview study (WP3).

Setting is community, comprised of employment settings in different sectors (public, private, third) in England, varying in size (small:10-49 workers; medium: 50-249 workers; large: >250 workers).

Sample size estimate: The aim is to recruit a minimum of 8 worksites ("clusters"), approximately 4 per arm. Up to 120 participants ("employees") will be recruited from these clusters over 12 months.

A nested interview study will be conducted, in which up to 40 people will be interviewed after 6 months. Participants in the interview study will include employees from the intervention arm, and stakeholders (identified by employees as having been involved in their support at work). Stakeholders may include line managers, company owners, human resources or occupational health specialists, or trade union representatives).

Organisations are randomised to either i) active control group (TAU: treatment as usual), or ii) TAU plus PAW Toolkit. Intervention participants can also opt in to receive up to 3 telephone calls with an occupational therapist. The content of the calls will include orientation to the PAW Toolkit and individually tailored advice on managing pain at work.

The following outcome measures will be collected (for detail, see Outcome Measures section):

A. Feasibility and acceptability outcomes:

B. Employer-reported outcome measures

C. Participant-reported outcome measures (PROMs)

ELIGIBILITY:
Inclusion Criteria (Organisations)

* organisations in England
* organisations with 10 or more employees.

Inclusion Criteria (Employee participants)

* working-age adults (employees)
* aged 18 and over
* self-reported chronic pain interfering with their ability to undertake or enjoy productive work
* able to comprehend English language
* able to provide informed consent.
* access to the internet to be able to access the web-based intervention and online surveys for data collection.

Exclusion Criteria (Organisations)

* organisations outside of England
* micro-organisations with fewer than 10 employees

Exclusion Criteria (Employee participants)

* unemployed at recruitment
* under 18 years of age
* no chronic pain at recruitment
* unable to comprehend English language
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Recruitment to the study | Baseline
  Number recruited to assess whether it would be possible to recruit to a definitive trial. The investigators will record the number recruited, characteristics of those recruited, and the timescale to recruit.
Acceptability of Intervention | 6 months
  Outcome to assess whether participants find the intervention acceptable. This will be self-reported in participant interviews at 6 months.
Fidelity of intervention (PAW Toolkit) | 3 months
  Intervention fidelity will be checked through collection of usage data for the PAW Toolkit, to assess engagement with the intervention. This data will be collected through a feedback form at 3 months.
Fidelity of intervention (OT support calls) | 3 months
  Intervention fidelity will be checked through recording of the uptake of occupational therapy support calls (to assess engagement with the intervention). This data will be collected through forms completed by the therapist at the time of each phone call which will be summed at 3 months.
Retention to the study at 3 months | 3 months
  Number of participants who complete the first follow-up outcome measures survey.
Retention to the study at 6 months | 6 months
  Number of participants who complete the second follow-up outcome measures survey.

SECONDARY OUTCOMES:
Work presenteeism | To assess change between time 0 (baseline), time 1 (3 months) and time 2 (6 months).
  Using the Work Limitations Questionnaire-25 (WLQ-25). To measure the degree to which pain interferes with specific components of job performance and the productivity impact of these work limitations. Scale range 0-111. Higher scores indicate worse outcome.
Work Ability | To assess change between time 0 (baseline), time 1 (3 months) and time 2 (6 months).
  Using the Work Ability Index Item1 (WAI1). Assesses current work ability compared to highest work ability ever. Scale range is 0-10. Higher scores indicate better outcome.
Work Self-Efficacy | To assess change between time 0 (baseline), time 1 (3 months) and time 2 (6 months).
  Using the Work Self-Efficacy Scale (WSES). This includes 10 items assessing perceptions regarding specific work domains such as the capability to manage interpersonal relationships (colleagues and direct superiors), to work with colleagues with different characteristics and experiences, to behave efficaciously in the work context, to learn new working methods, to respect schedules and work deadlines, and to achieve assigned goals. Respondent rates capability on each item from 1 (Not well at all) to 5 (Very well). Higher score indicates better outcome.
Job satisfaction | To assess change between time 0 (baseline), time 1 (3 months) and time 2 (6 months).
  Global single-item measure. Using the item: 'Taking everything into consideration, how do you feel about your job as a whole?' with responses ranging from 1 = extremely dissatisfied through to 5 = extremely satisfied. Higher score indicates better outcome.
Job stressfulness | To assess change between time 0 (baseline), time 1 (3 months) and time 2 (6 months).
  Global single-item measure. Using the item: 'In general, how stressful do you find your job?' with responses on a 5 point scale ranging from 1 = 'not at all stressful' through to 5 = 'extremely stressful'. Higher score indicates worse outcome.
Turnover intentions | To assess change between time 0 (baseline), time 1 (3 months) and time 2 (6 months).
  Global single item measure. Using the item: 'Are you considering leaving your job due to your pain?' (yes or no). Negative response is better outcome.
Depression | To assess change between time 0 (baseline), time 1 (3 months) and time 2 (6 months).
  Using the Patient Health Questionnaire (PHQ-2). Scale is used to screen for depression. Scores ranges from 0-6. Higher scores indicate worse outcome.
Anxiety | To assess change between time 0 (baseline), time 1 (3 months) and time 2 (6 months).
  Using the General Anxiety Disorder (GAD-7). Used as a screening tool and severity measure for generalised anxiety disorder. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Total score ranges from 0-21. Higher scores indicate worse outcome.
Health-related quality of life | To assess change between time 0 (baseline), time 1 (3 months) and time 2 (6 months).
  Using the EuroQol Five Dimensions Questionnaire (EQ-5D-5L). Comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. For instance, 'slight problems' (e.g. 'I have slight problems in walking about') is always coded as '2'. The digits for the five dimensions can be combined in a 5-digit code that describes the respondent's health state. Higher scores indicate worse outcome.
Impairments in work and activities | To assess change between time 0 (baseline), time 1 (3 months) and time 2 (6 months).
  Using the Work Productivity and Impairments Scale (WPAI-GH). Measures impairments in both paid work and unpaid work. It measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. The WPAI yields four types of scores:
  1. Absenteeism (work time missed); 2. Presenteeism (impairment at work / reduced on-the-job effectiveness); 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism); 4. Activity Impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity (worse outcomes).
Health resource use questionnaire | Cumulative health resource use at time 0 (baseline), time 1 (3 months), time 2 (6 months)
  Using a health care resource use questionnaire to measure completion rates for items of resource use, such as frequency of use of secondary and primary care, social care, private health care, and medications. Items are adapted from health economics data capture in previous research with pain populations. Minimum score zero, no maximum. Higher scores indicate greater frequency of resource use.
Social support at work | To assess change between time 0 (baseline), time 1 (3 months) and time 2 (6 months).
  Using the Demand Control Support Questionnaire (DCSQ) - Social Support Sub-Scale consisting of 6 items covering: pleasant atmosphere, spirit of unity, colleagues support, helpful colleagues, relationship with superiors, relationship with colleagues. Respondents are asked to report their levels of agreement or disagreement on a four-point Likert scale. Higher values indicate better outcome (higher social support at work, score range 6-24).

OTHER OUTCOMES:
Organisation-reported sickness absence records | To assess change between time 0 (baseline), time 1 (3 months) and time 2 (6 months).
  Organisational records of sickness absence rates for participating employees.
Employment status | To document any changes in participant's employment status between time 0 (baseline), time 1 (3 months) and time 2 (6 months).
  Using items from the Work Transitions Index (WTI) covering employment status, occupation and working hours.
Nature of work | To document any changes in participant's nature of work between time 0 (baseline), time 1 (3 months) and time 2 (6 months).
  Using UK Standard Job Skill Classification (Job Skill Level 1-4): Main job title and industry working in.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Blake, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Protocol - details shared via clinical trials.gov and protocol manuscript (with informed consent form) to be submitted to an open access peer-reviewed journal within 6 months.
  Data Management Plan will be publicly available on https://dmponline.dcc.ac.uk prior to study start.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Protocol - baseline (registration) 6 months (submitted protocol for publication) Statistical analysis plan - baseline Informed consent form - 6 months (submitted protocol for publication)
Access Criteria: Protocol - details shared via clinical trials.gov and protocol manuscript (with informed consent form) to be submitted to an open access peer-reviewed journal within 6 months.
  Data Management Plan will be publicly available on https://dmponline.dcc.ac.uk prior to ethical approval and study start.
URL: https://dmponline.dcc.ac.uk

REFERENCES:
- [Background] Blake H, Somerset S, Greaves S. The Pain at Work Toolkit for Employees with Chronic or Persistent Pain: A Collaborative-Participatory Study. Healthcare (Basel). 2021 Dec 29;10(1):56. doi: 10.3390/healthcare10010056. PMID 35052220
- [Background] Blake H, Chaplin WJ, Wainwright E, Taylor G, McNamee P, McWilliams D, Abbott-Fleming V, Holmes J, Fecowycz A, Walsh DA, Walker-Bone K. The Web-Based Pain-at-Work Toolkit With Telephone Support for Employees With Chronic or Persistent Pain: Protocol for a Cluster Randomized Feasibility Trial. JMIR Res Protoc. 2023 Oct 30;12:e51474. doi: 10.2196/51474. PMID 37902814
- [Derived] Blake H, Abbott-Fleming V, Greaves S, Somerset S, Chaplin WJ, Wainwright E, Walker-Bone K. Five years of patient and public involvement and engagement (PPIE) in the development and evaluation of the Pain-at-Work toolkit to support employees' self-management of chronic pain at work. Res Involv Engagem. 2025 Jul 15;11(1):81. doi: 10.1186/s40900-025-00757-5. PMID 40665420
- See also: Nuffield Foundation and Arthritis UK Research Funding (Award Ref: OBF/FR-000023820) — https://www.nuffieldfoundation.org/project/the-paw-trial-feasibility-and-acceptability-of-the-pain-at-work-toolkit